CLINICAL TRIAL: NCT06591286
Title: Effects of Real-time Continuous Glucose Monitoring System on Hospital-to-home Transitional Blood Glucose Control and Self-efficacy Among Patients With Type 2 Diabetes Treated With Insulin
Brief Title: Effects of Real-time Continuous Glucose Monitoring System on Hospital-to-home Transitional Blood Glucose Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Professor, Chief Physician, Deputy Director, Department of Endocrinology and Metabolism, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT20240903
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Continuous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group (75 cases) will wear real-time CGM to monitor blood glucose for 12 weeks, followed by 36 weeks of follow-up.
  Interventions: Device: RT-CGM
- Control group (Other): The control group (75 cases) is self-monitored by traditional SMBG for 12 weeks at a frequency of no less than 4 times a week, followed by 36 weeks of follow-up.
  Interventions: Device: SMBG

INTERVENTIONS:
Device: RT-CGM — This group of patients will wear RT-CGM for blood glucose monitoring for three months.
  Arms: Intervention group
Device: SMBG — This group of patients will use a a fingertip glucose meter for blood glucose monitoring for three months, and the monitoring frequency was not less than 4 times per week.
  Arms: Control group

SUMMARY:
Glucose monitoring is an important part of self-management for patients with diabetes. The results of glucose monitoring not only help to assess the degree of glucose metabolism disorders in patients, but also help physicians to make clinical decisions and guide patients in self-management. Despite extensive efforts and advances in diabetes management during hospitalization, glucose control after patients is discharged home remains a challenge. This trial aims to explore the effect of real-time continuous glucose monitoring (RT-CGM) system compared to self-monitoring of blood glucose (SMBG) group on glucose and self-efficacy of type 2 diabetes patients treated with insulin after discharge from the hospital.

DETAILED DESCRIPTION:
Glycemic management of patients with diabetes after discharge home is extremely challenging, especially for those requiring insulin therapy. The use of a real-time continuous glucose monitoring (RT-CGM) system may improve glycemic control and self-efficacy in patients with type 2 diabetes treated with insulin after discharge from the hospital.

One hundred and fifty insulin-treated adults with type 2 diabetes were randomly assigned to receive either RT-CGM or self-monitoring of blood glucose (SMBG) at hospital discharge for a 12-week monitoring intervention and a 36-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 80 years old.
2. Type 2 diabetes admitted to Department of Endocrinology and Metabolism.
3. 8% ≤ HbA1c ≤ 12% in the last 1 month.
4. Insulin therapy within 1 month of planned discharge from hospital.
5. Frequency of self-monitoring of blood glucose <4 times per week and no use of real-time continuous glucose monitoring system in the 3 months prior to hospitalisation.
6. Willing and able to provide written informed consent and comply with the requirements of this study.

Exclusion Criteria:

1. Oral steroid hormone therapy.
2. Patients with acute complications of diabetes (including Diabetic ketoacidosis, hyperglycemia and hyperosmolality, Lactic acidosis)
3. Patients with severe liver disease (alanine aminotransferase or glutamine aminotransferase exceeding more than three times the upper limit of normal).
4. Patients with severe kidney injury or end-stage renal disease (eGFR < 30 mL/min/1.73 m2).
5. Participants were unable to tolerate tape adhesive around sensor placement area, or with medically documented allergy towards the adhesive (glue) of plasters, or with serious skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) around sensor placement area.
6. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
7. Pregnant, breastfeeding, women of childbearing age who are unwilling to use contraception during the study period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Time in range (3.9~10.0mmol/L, %) | 12 weeks
  Percentage of time within glucose level of 3.9-10.0 mmol/L (70-180 mg/dL) measured by CGM.

SECONDARY OUTCOMES:
HbA1c (%) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Glycated hemoglobin (%)
Time in range (3.9~10.0mmol/L, %) | 4weeks, 8weeks, 24weeks, 48 weeks
  Percentage of time within glucose level of 3.9-10.0 mmol/L (70-180 mg/dL) measured by CGM.
Time above range (>10.0mmol/L, %) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Percentage of time above glucose level of 10.0 mmol/L (180 mg/dL) measured by CGM.
Time below range (<3.9mmol/L, %) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Percentage of time below glucose level of 3.9 mmol/L (70 mg/dL) measured by CGM.
Coefficient of variation (CV) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Standard deviation divided by mean glucose level measured by CGM.
Standard deviation (SD) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Standard deviation of blood glucose measurements during CGM.
Mean amplitude of glycemic excursions (MAGE) | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  Mean amplitude of glycemic excursions (MAGE) is the average value of all amplitude of glycemic excursions.
Diabetes management self-efficacy | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  The Chinese version of Diabetes Management Self-efficacy Scale (DMSES) is used to evaluate the patients' self-efficacy
Diabetes Self Care Activities | 4weeks, 8weeks, 12 weeks, 24weeks, 48weeks
  The Chinese version of Summary of Diabetes Self Care Activities (SDSCA) is used to evaluate the patients' self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Dr., Principal Investigator — Shanghai 6th People's Hospital
Locations (1):
- Shanghai 6th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No